CLINICAL TRIAL: NCT03851159
Title: Nyaditum Resae® (a Food Supplement) as a Co-adjuvant During First-line Treatment for Active Pulmonary Tuberculosis and Its Impact on the Gut Microbiota - a Pilot Double-blind Randomised Controlled Trial
Brief Title: Nyaditum Resae® as a Co-adjuvant During Treatment for Active Pulmonary Tuberculosis and Its Impact on the Gut Microbiota
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Principal Investigator, Grant Theron, Associate Professor, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: N14_10_136
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis
Keywords: Microbiome
MeSH Terms: conditions — Tuberculosis | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Intervention: HIV-negative (Placebo Comparator): HIV-negative patients are selected to receive the placebo for the first two weeks of first-line TB treatment.
  Interventions: Other: Mannitol
- Intervention: HIV- (Experimental): HIV-negative patients are selected to receive the food supplement for the first two weeks of first-line TB treatment.
  Interventions: Dietary Supplement: Nyaditum resae®
- No Intervention: HIV+ (Placebo Comparator): HIV-positive patients are selected to receive the placebo for the first two weeks of first-line TB treatment.
  Interventions: Other: Mannitol
- Intervention: HIV+: (Experimental): HIV-positive patients are selected to receive the food supplement for the first two weeks of first-line TB treatment.
  Interventions: Dietary Supplement: Nyaditum resae®

INTERVENTIONS:
Dietary Supplement: Nyaditum resae® — Heat-killed Mycobacterium manresensis
  Arms: Intervention: HIV+:; Intervention: HIV-
Other: Mannitol — Placebo
  Arms: No Intervention: HIV+; No Intervention: HIV-negative

SUMMARY:
This will be the first study to evaluate the use of Nyaditum resae® as a potential agent for reducing antibiotic-associated gut dysbiosis in patients with drug-susceptible TB, and potentially improving clinical and microbiological markers of outcome

DETAILED DESCRIPTION:
About one tenth of the 1.7 billion individuals infected with Mycobacterium tuberculosis (Mtb) will progress to active tuberculosis (TB). This probability increases in people with human immunodeficiency virus (HIV) and other risk co-morbidities such as malnutrition, diabetes and substance abuse. Chronic microbial colonisation with unrelated bacteria are associated with TB pathogenesis (e.g., mice colonised with Helicobacter hepaticus exhibit poor control of TB), indicating that the gut microbiota may modulate progression to active TB. Furthermore, first-line TB treatment (Isoniazid, Rifampicin, Ethambutol, Pyrazinamide; HREZ) depletes gut commensal bacteria (Ruminococcus, Coprococcus and Bifidobacterium) with immunomodulatory roles [interleukin (IL)-1, interferon (IFN)-γ and Th17 responses, respectively).

Recent work identified heat-killed Mycobacterium manresensis (hkMm), a harmless member of the fortuitum complex naturally found in drinking water, as a promising candidate for reducing the risk of active TB. Mtb-infected mice treated with hkMm had significantly reduced lung pathology (fewer and smaller lesions,) bacillary load and proinflammatory cytokines (TNF-α, IFN-γ, IL-6, and IL-17) compared to untreated control mice, and in mice receiving hkMm with HREZ, survival rates were significantly increased. Moreover, mice treated with hkMm had increased microbial diversity and an altered gut microbial composition relative to untreated mice. This could prove beneficial for TB patients during prolonged antibiotic treatment as supplementation with hkMm may help protect gut microbiota, and potentially improve clinical outcome.

In individuals with and without latent M. tuberculosis infection, two weeks of daily oral doses of Nyaditum resae® (a preparation of hkMm approved as a food supplement by Manremyc) demonstrated enhanced effector and memory specific regulatory T-cell responses. Similar clinical trials with Nyaditum resae® are currently being done in paediatrics (NCT02581579) and close contacts of active TB cases in Tbilisi, Georgia (NCT02897180; 2017-2023). The probiotic is also being registered as a food supplement in several countries.

In the proposed study, the efficacy of Nyaditum resae® in reducing antibiotic-associated gut dysbiosis and disease progression in patients with active TB will be tested. To do this, the investigators will assess changes in the microbiota during treatment (with or without Nyaditum resae® supplementation) and attempt to identify genera associated with a favourable or unfavourable treatment outcome in TB patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* New cases
* Sputum Xpert Ultra (Xpert) positive for Mycobacterium tuberculosis
* Have not initiated TB treatment
* If HIV-positive, are stable on antiretroviral therapy

Exclusion Criteria:

* Resistance to any of the first-line drugs (Xpert rifampicin-resistant)
* Previous TB
* Diabetes mellitus
* Taking immunomodulatory drugs (e.g. cancer chemotherapy, tumour necrosis factor (TNF) inhibitors or other anti-inflammatory medication, phosphodiesterase inhibitors, corticosteroids within the past 6 months, and cholesterol-lowering drugs)
* Pregnant or lactating women
* Chronic hepatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome composition in placebo versus experimental arm | Up to 18 months
  Gut microbial composition determined by next-generation sequencing of bacterial DNA in stool

SECONDARY OUTCOMES:
Cytokine and cluster of differentiation (CD)4+ T-cell response in placebo versus experimental arm | Up to 18 months
  Cytokines responses profiled using commercial human cytokine panel, and T-cell responses characterised by flow cytometry on isolated peripheral blood mononuclear cells
Time to sputum conversion and reduction in bacillary load | Up to 6 months
  Culture used to assess sputum conversion and bacillary load

CONTACTS AND LOCATIONS:
Overall Officials: Grant Theron, PHD, Principal Investigator — University of Stellenbosch
Locations (2):
- South Africa (2):
  - Scottsdene Clinic, Cape Town, Western Cape
  - Wallacedene Clinic, Cape Town, Western Cape